CLINICAL TRIAL: NCT01146431
Title: Memory During Inhalation Anesthesia Performed With or Without Bispectral Index (BIS) in Patients Undergoing Thyroidectomy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Catholic University of the Sacred Heart (Other)
Responsible Party: Catholic University of Sacred Heart, Catholic University of Sacred Heart
Other Study IDs: A/1051/2009
Record Dates: First submitted 2010-06-09; First posted 2010-06-17 (Estimated); Last update posted 2011-02-09 (Estimated); Status verified 2010-01

CONDITIONS: Thyroidectomy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

GROUPS / COHORTS (2):
- Hemodynamic parameters: Hemodynamic parameters will be used as a guide for anesthesia.
  Interventions: Drug: Inhaled anesthetics
- BIS: Bispectral Index (BIS) will be used as a guide for anesthesia.
  Interventions: Drug: Inhaled anesthetics

INTERVENTIONS:
Drug: Inhaled anesthetics — Inhaled anaesthetic drugs (sevoflurane or desflurane) concentration will be changed on the basis of hemodynamic parameters (mean arterial pressure and heart rate greater or less than 20% compared to preoperative values).
  Groups: Hemodynamic parameters
Drug: Inhaled anesthetics — Inhaled anaesthetic drugs (sevoflurane or desflurane) concentration will be changed on the basis of Bispectral Index (BIS) value which will be maintained between 40 and 50.
  Groups: BIS

SUMMARY:
The purpose of this study is 1) to investigate whether the use of BIS as a guide to the administration of inhaled anesthetic (sevoflurane or desflurane) compared with the use of hemodynamic parameters (blood pressure and heart rate) would affect the occurrence of implicit memory and /or dreams recall and 2) to check whether the occurrence of implicit memory and/or dreams recall is related with MAC (Minimal Alveolar Concentration) of inhalational anesthetics and/or preoperative anxiety levels.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 70 years
* Class-ASA Physical Status I-II

Exclusion Criteria:

* Psychiatric or neurological disorders and/or hearing disorders
* Obesity (Body Mass Index > 30)
* Drug addiction, alcoholism
* Patient with difficulty in understanding italian language and/or education level below middle school

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing general anesthesia for thyroidectomy
Sampling Method: Probability Sample
Enrollment: 130 (Estimated)
Dates: Start 2010-06

PRIMARY OUTCOMES:
Implicit memory | Approximately 24 hours after surgery
  Implicit memory will be investigated using free association test: patients, during maintenance of anesthesia, will listen a piece of one of two stories, "Puss in Boots" or "Pinocchio", each followed by four keywords. Approximately 24 hours after surgery, patients will be asked to associate the first thing that comes to mind with these keywords in order to highlight the presence of implicit memory. The test will be repeated twice and will be positive if the patient will reply with the title of the story or a word of it.

SECONDARY OUTCOMES:
Dreams recall | Approximately 5 minutes after awakening from anesthesia
  A first interview about dreams recall will be carried out 5 minutes after awakening from anesthesia. Patients will be asked about dream content.
Explicit memory | Approximately 24 hours after surgery
  Patients will be asked about the last thing they remembered before going to sleep; the first thing they remember when they woke up; and anything which happen in between, including sounds, dreams and imagination.
Dreams recall | Approximately 24 hours after anaesthesia
  Patients will be asked again about dreams recall. The content of dreams will be analyzed using the 5-point Likert scales which contains the following dreams characteristics: memory content, emotional content, emotional intensity, vivid description, amount of sounds, meaning, how much movement, strange, episodic content, references to episodes of life.

CONTACTS AND LOCATIONS:
Locations (1):
- Catholic University of Sacred Heart, Rome, Italy, Italy